CLINICAL TRIAL: NCT03699124
Title: A Randomized, Double-blind, Multicenter Phase III Trial to Evaluate Immunogenicity and Safety of Three Consecutive Production Lots of a Freeze-dried Formulation of MVA-BN® Smallpox Vaccine in Healthy, Vaccinia-naïve Subjects
Brief Title: Freeze-Dried MVA-BN® Lot Consistency Smallpox Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POX-MVA-031
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2020-07

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GP 1: two doses of FD MVA-BN--Lot 1 (Active Comparator): Healthy, vaccinia-naïve subjects receiving two subcutaneous (SC) vaccinations, four weeks apart with freeze-dried (FD) MVA-BN® - Lot 1
  Interventions: Biological: FD MVA-BN
- GP 2: two doses of FD MVA-BN--Lot 2 (Active Comparator): Healthy, vaccinia-naïve subjects receiving two subcutaneous (SC) vaccinations, four weeks apart with freeze-dried (FD) MVA-BN® - Lot 2
  Interventions: Biological: FD MVA-BN
- GP 3: two doses of FD MVA-BN--Lot 3 (Active Comparator): Healthy, vaccinia-naïve subjects receiving two subcutaneous (SC) vaccinations, four weeks apart with freeze-dried (FD) MVA-BN® - Lot 3
  Interventions: Biological: FD MVA-BN

INTERVENTIONS:
Biological: FD MVA-BN — Vaccinations with a 0.5 mL dose of vaccine containing at least 0.5 x 10E8 Infectious Units (Inf.U)

SUMMARY:
This is a Phase 3 multicenter trial to evaluate safety and immune response of three consecutive production lots of freeze-dried (FD) MVA-BN smallpox vaccine. The vaccine will be given to healthy subjects who do not have a smallpox scar.

Approximately 1110 subjects will be randomly enrolled into one of three groups:

Group 1 will include 370 subjects, who will receive two separate injections (shot) with a short needle, given below the skin of the upper arm with 0.5 mL FD MVA-BN (Lot 1).

Group 2 will include 370 subjects, who will receive two separate injections (shot) with a short needle, given below the skin of the upper arm with 0.5 mL FD MVA-BN (Lot 2).

Group 3 will include 370 subjects, who will receive two separate injections (shot) with a short needle, given below the skin of the upper arm with 0.5 mL FD MVA-BN (Lot 3).

The primary objective of the trial is to show that the immune response elicited (produced) by three consecutively produced MVA-BN lots are statistically (numerically) comparable.

ELIGIBILITY:
Inclusion Criteria:

* The subject has read, signed and dated the ICF
* Body Mass Index ≥ 18.5 and < 35
* Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal (defined as ≥ 12 months without a menstrual period) or surgically sterilized. Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products).
* WOCBP must have a negative serum pregnancy test at screening (please note: a negative urine pregnancy test is required within 24 hours prior to each vaccination)
* White blood cells ≥ 2500/mm3 < ULN (Upper Limit of Normal)
* Absolute neutrophil count (ANC) within normal limits
* Hemoglobin within normal limits
* Platelets within normal limits
* Adequate renal function defined as a calculated Creatinine Clearance (CrCl) > 60 mL/min as estimated by the Cockcroft-Gault equation: (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min). For women the result, calculated with the above formula, has to be multiplied by 0.85 = CrCl (mL/min)
* Adequate hepatic function defined as: Total bilirubin ≤ 1.5 x ULN in the absence of other evidence of significant liver disease Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 1.5 x ULN
* Electrocardiogram (ECG) without clinically significant findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions in a row, ST elevation consistent with ischemia).

Exclusion Criteria:

* Typical vaccinia scar
* Known or suspected history of smallpox vaccination
* History of vaccination with any poxvirus-based vaccine
* US Military service prior to 1991 or after January 2003
* Pregnant or breast-feeding women
* Uncontrolled serious infection, i.e. not responding to antimicrobial therapy
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or would limit the subject's ability to complete the trial
* History of or active autoimmune disease, persons with vitiligo or thyroid disease taking thyroid replacement are not excluded
* Known or suspected impairment of immunologic function including, but not limited to, human immunodeficiency virus (HIV) Infection, clinically significant liver disease (including chronic active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection), diabetes mellitus
* History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site.
* History or clinical manifestation of clinically significant and severe hematological, pulmonary, central nervous, cardiovascular or gastrointestinal disorders
* Clinically significant mental disorder not adequately controlled by medical treatment
* History of coronary heart disease, myocardial infarction, angina pectoris, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor
* Abnormal Troponin I level > ULN
* Known history of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before age 50 years
* Active or history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the past 6 months)
* Known allergy to MVA-BN vaccine or any of its constituents, e.g. tris (hydroxymethyl)-amino methane, including known allergy to egg or aminoglycosides
* History of anaphylaxis or severe allergic reaction to any vaccine
* Acute disease (illness with or without a fever) at the time enrollment
* Body temperature ≥ 100.4°F (≥ 38.0°C) at the time of enrollment
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to or after trial vaccination
* Having received any vaccinations or planned vaccinations with a killed/inactivated vaccine within 14 days prior to or after trial vaccination
* Chronic systemic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (Visit 5)
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (Visit 5)
* Use of any investigational or non-registered product within 30 days preceding the first dose of the trial vaccine, or planned administration of such a drug during the trial period
* Trial personnel

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1129 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar T Overton, MD, Principal Investigator — University of Alabama at Birmingham
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Optimal Research, LLC (Synexus), Melbourne, Florida
  - Optimal Research, LLC (Synexus), Peoria, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky Healthcare Chandler Hospital, Lexington, Kentucky
  - Optimal Research, LLC (Synexus), Rockville, Maryland
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner Overton E, Schmidt D, Vidojkovic S, Menius E, Nopora K, Maclennan J, Weidenthaler H. A randomized phase 3 trial to assess the immunogenicity and safety of 3 consecutively produced lots of freeze-dried MVA-BN(R) vaccine in healthy adults. Vaccine. 2023 Jan 9;41(2):397-406. doi: 10.1016/j.vaccine.2022.10.056. Epub 2022 Nov 29. PMID 36460535

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Started (Randomized) | 377 | 375 | 377
Completed (Active study period) | 332 | 335 | 337
Not Completed | 45 | 40 | 40
Not completed — Adverse Event | 6 | 5 | 2
Not completed — Death | 0 | 2 | 0
Not completed — Lost to Follow-up | 20 | 16 | 15
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 14 | 13
Not completed — Other reasons | 5 | 3 | 10

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all subjects who were randomized and received at least one dose of trial vaccine, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3 | Total
Number analyzed (Participants) | 377 | 375 | 377 | 1129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 377 | 375 | 377 | 1129
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (7.31) | 30.6 (7.29) | 30.7 (7.50) | 30.7 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 213 | 207 | 630
  Male | 167 | 162 | 170 | 499
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 20 | 25 | 73
  Not Hispanic or Latino | 348 | 354 | 349 | 1051
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4 | 8
  Asian | 17 | 13 | 13 | 43
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 58 | 55 | 59 | 172
  White | 292 | 295 | 293 | 880
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 377 | 375 | 377 | 1129

OUTCOME MEASURES:

1. Primary Outcome: Vaccinia-Specific Neutralizing Antibodies Measured by Plaque Reduction Neutralization Test (PRNT)
Description: Vaccinia-specific neutralizing antibody titers below the lower limit of quantitation are given a value 10, i.e., half of the PRNT lower limit of quantitation of 20.
Time Frame: Two weeks post second vaccination; approximately Week 6.
Population: The Per Protocol Set includes all randomized subjects who received at least one vaccination and had no major protocol deviations that might have a substantial impact on the immunogenicity results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 327 | 331 | 330
Titer | 252.7 [231.3 to 276.0] | 269.9 [243.2 to 299.7] | 242.0 [219.5 to 266.8]
Statistical Analysis 1: Comparison: GP 1: Two Doses of FD MVA-BN--Lot 1 vs GP 2: Two Doses of FD MVA-BN--Lot 2; Test type: Equivalence — Equivalence between two lot groups is demonstrated if the confidence interval of the ratio of the GMTs lies within the interval [½, 2]. For the trial to be successful, all three lot group comparisons must be equivalent by this definition; GMT Ratio = 0.936, 95% CI 2-sided [0.816 to 1.073]
Statistical Analysis 2: Comparison: GP 2: Two Doses of FD MVA-BN--Lot 2 vs GP 3: Two Doses of FD MVA-BN--Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.115, 95% CI 2-sided [0.967 to 1.287]
Statistical Analysis 3: Comparison: GP 1: Two Doses of FD MVA-BN--Lot 1 vs GP 3: Two Doses of FD MVA-BN--Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.044, 95% CI 2-sided [0.915 to 1.191]

2. Secondary Outcome: Vaccinia-Specific Total Antibodies Measured by Enzyme-Linked Immunosorbant Assay (ELISA)
Description: Vaccinia-specific total antibody titers below the lower limit of quantitation are given a value 100, i.e., half of the ELISA lower limit of quantitation of 200.
Time Frame: Two weeks post second vaccination; approximately Week 6.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 327 | 331 | 330
Titer | 1222 [1123.3 to 1329.4] | 1311 [1195.7 to 1437.5] | 1226.1 [1118.1 to 1344.6]

3. Secondary Outcome: Seroconversion Rates for Vaccinia-Specific Neutralizing Antibodies by PRNT
Description: Seroconversion is defined as either the appearance of antibody titers >= LLOQ for subjects with a titer below LLOQ at baseline, or a doubling (or more) of the antibody titer compared to the baseline titer for subjects with a titer equal or above the LLOQ at baseline. The LLOQ for PRNT is 20.
Time Frame: Two weeks post second vaccination; approximately Week 6.
Population: The Per Protocol Set includes all randomized subjects who received at least one vaccination and had no major protocol deviations that might have a substantial impact on the immunogenicity results. Only subjects who had both a baseline and two weeks post second vaccination titer results are included.
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 326 | 331 | 330
Participants | 325 | 328 | 327

4. Secondary Outcome: Seroconversion Rates for Vaccinia-Specific Total Antibodies by ELISA
Description: Seroconversion is defined as either the appearance of antibody titers >= LLOQ for subjects with a titer below LLOQ at baseline, or a doubling (or more) of the antibody titer compared to the baseline titer for subjects with a titer equal or above the LLOQ at baseline. The LLOQ for ELISA is 200.
Time Frame: Two weeks post second vaccination; approximately Week 6.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 326 | 331 | 330
Participants | 323 | 325 | 326

5. Secondary Outcome: Pearson Correlation Coefficient Between the log10 Transformed PRNT Titers and the log10 Transformed ELISA Titers
Description: Pearson correlation coefficient calculated on the log10 PRNT vs. ELISA titers at 2 weeks post second vaccination.
Time Frame: Two weeks post second vaccination; approximately Week 6.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 327 | 331 | 330
Correlation Coefficient | 0.657 [0.5901 to 0.7142] | 0.657 [0.5910 to 0.7142] | 0.656 [0.5893 to 0.7131]

6. Secondary Outcome: Occurrence, Relationship and Intensity of Any Serious Adverse Event (SAE) at Any Time During the Trial
Description: Occurrence is defined as the number of participants who experienced an SAE. Related SAEs are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, published September 2007, where >= Grade 3 is either Severe or Potentially Life Threatening.
Time Frame: Overall study, ie from first vaccination at Visit 1 through the Follow-up Visit approximately 32 weeks post first vaccination.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants
  Any Serious Adverse Event | 1 | 7 | 1
  Related Serious Adverse Event | 0 | 0 | 0
  Serious Adverse Event >= Grade 3 | 0 | 5 | 1

7. Secondary Outcome: Occurrence, Relationship and Intensity of Any Cardiac Sign or Symptom Indicating a Case of Myo-/Pericarditis at Any Time During the Trial.
Description: Occurrence is defined as the number of participants who experienced an event falling in the system organ class of "Cardiac disorders" per MedDRA version 22.0. Related cardiac signs and symptoms are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, published September 2007, where >= Grade 3 is either Severe or Potentially Life Threatening.
Time Frame: as for outcome 6
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants
  Any Cardiac Sign or Symptom | 1 | 2 | 1
  Any Related Cardiac Sign or Symptom | 0 | 0 | 0
  Any Cardiac Sign or Symptom >=Grade 3 | 0 | 0 | 0

8. Secondary Outcome: Occurrence of Any Grade 3 or 4 Unsolicited AEs Probably, Possibly or Definitely Related to the Trial Vaccine
Description: Related AEs are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, published September 2007, where Grade 3 is Severe and Grade 4 is Potentially Life Threatening.
Time Frame: Within 28 days (and up to 35 days) after each vaccination, ie, from Visit 1 to Visit 3 for the first vaccination and from Visit 3 to Visit 5 for the second vaccination based on the protocol scheduled visits.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants | 2 | 0 | 1

9. Secondary Outcome: Occurrence, Relationship and Intensity of Unsolicited AEs
Description: Occurrence is defined as the number of participants who experienced an unsolicited AE. Related unsolicited AEs are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials, published September 2007, where >= Grade 3 is either Severe or Potentially Life Threatening.
Time Frame: as for outcome 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants
  Any Unsolicited AE | 88 | 110 | 98
  Any Related Unsolicited AE | 33 | 38 | 37
  Any Unsolicited AE >= Grade 3 | 6 | 8 | 7

10. Secondary Outcome: Occurrence and Intensity of Solicited Local AEs (Redness, Swelling, Induration, Pruritus and Pain).
Description: Occurrence is defined as the number of participants who experienced a solicited local AE. Intensity is defined per the protocol for each local event type. For injection site erythema, swelling, and induration the intensity is graded based on the maximum diameter as Grade 1: < 30mm, Grade 2: >= 30 - < 100mm, Grade 3: >= 100mm. Intensity for pruritis is defined as Grade 1: mild, Grade 2: moderate, Grade 3: severe. Intensity for injection site pain is defined as Grade 1: Painful on touch, Grade 2: Painful when moving the limb, Grade 3: Spontaneously painful/prevents normal activity. If a participant experienced the local event after both vaccinations, the maximum intensity is presented.
Time Frame: During the 8 day period (day of vaccination and the following 7 days) after each vaccination, ie Days 1-8 for the first vaccination and Days 28-35 for the second vaccination based on the protocol scheduled visits.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants
  Any Solicited Local AEs | 338 | 348 | 344
  Any Redness | 271 | 283 | 272
  Redness Grade 1 | 84 | 110 | 87
  Redness Grade 2 | 143 | 131 | 156
  Redness Grade 3 | 44 | 42 | 29
  Any Swelling | 215 | 233 | 236
  Swelling Grade 1 | 88 | 121 | 118
  Swelling Grade 2 | 110 | 87 | 106
  Swelling Grade 3 | 17 | 25 | 12
  Any Induration | 215 | 226 | 229
  Induration Grade 1 | 98 | 126 | 123
  Induration Grade 2 | 106 | 92 | 100
  Induration Grade 3 | 11 | 8 | 6
  Any Pruritis | 210 | 230 | 198
  Pruritis Grade 1 | 160 | 181 | 159
  Pruritis Grade 2 | 40 | 42 | 29
  Pruritis Grade 3 | 10 | 7 | 10
  Any Injection Site Pain | 325 | 330 | 329
  Injection Site Pain Grade 1 | 118 | 112 | 124
  Injection Site Pain Grade 2 | 161 | 173 | 162
  Injection Site Pain Grade 3 | 46 | 45 | 43

11. Secondary Outcome: Duration of Solicited Local AEs (Redness, Swelling, Induration, Pruritus and Pain).
Description: Number of days from the start of the local event to resolution. If a participant experienced the local event after both vaccinations, the longer duration is presented. Subjects who had a missing resolution date for the event are not included in the analysis.
Time Frame: Starting during the 8 day period (day of vaccination and the following 7 days) after each vaccination, ie, Days 1-8 for the first vaccination and Days 28-35 for the second vaccination based on the protocol scheduled visits, through resolution.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Days
  Redness: number analyzed (Participants) | 271 | 283 | 272
  Redness | 7.1 (6.53) | 6.5 (5.06) | 6.6 (5.39)
  Swelling: number analyzed (Participants) | 215 | 233 | 236
  Swelling | 6.7 (6.47) | 6 (5.04) | 5.9 (4.52)
  Induration: number analyzed (Participants) | 213 | 226 | 227
  Induration | 18 (24.04) | 13.9 (13.12) | 15 (15.01)
  Pruritis: number analyzed (Participants) | 210 | 230 | 198
  Pruritis | 5 (5.7) | 4.4 (3.24) | 4.4 (3.87)
  Pain: number analyzed (Participants) | 325 | 330 | 329
  Pain | 6.9 (4.41) | 7.1 (4.44) | 6.7 (3.64)

12. Secondary Outcome: Occurrence, Relationship, and Intensity of Solicited General AEs (Pyrexia, Headache, Myalgia, Nausea, Fatigue and Chills).
Description: Occurrence is defined as the number of participants who experienced a solicited general AE. Related solicited general AEs are defined as those for which causality to trial vaccine was considered possible, probable, definite, or was missing. Intensity is defined per the protocol for each general event type. For pyrexia (increased body temperature) grading is defined as Grade 1: ≥ 99.5 - < 100.4°F (≥ 37.5 - < 38.0°C), Grade 2:≥ 100.4 - < 102.2°F (≥ 38.0 - < 39.0°C), Grade 3:≥ 102.2 - < 104°F (≥ 39.0 - < 40.0°C), and Grade 4: ≥ 104°F (≥ 40.0°C). Intensity for headache, myalgia, nausea, fatigue and chills is defined as Grade 1: mild, Grade 2: moderate, Grade 3: severe. If a participant experienced the general event after both vaccinations, the maximum intensity is presented.
Time Frame: as for outcome 10
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Participants
  Any Solicited General AEs | 253 | 267 | 266
  Any Related Solicited General AEs | 246 | 256 | 252
  Any Pyrexia | 47 | 60 | 63
  Pyrexia Grade 1 | 39 | 48 | 49
  Pyrexia Grade 2 | 7 | 8 | 13
  Pyrexia Grade 3 | 1 | 4 | 1
  Pyrexia Grade 4 | 0 | 0 | 0
  Any Related Pyrexia | 47 | 57 | 55
  Any Headache | 146 | 157 | 155
  Headache Grade 1 | 96 | 102 | 120
  Headache Grade 2 | 36 | 44 | 25
  Headache Grade 3 | 14 | 11 | 10
  Any Related Headache | 140 | 145 | 145
  Any Myalgia | 166 | 173 | 175
  Myalgia Grade 1 | 115 | 116 | 116
  Myalgia Grade 2 | 38 | 47 | 39
  Myalgia Grade 3 | 13 | 10 | 20
  Any Related Myalgia | 159 | 167 | 167
  Any Nausea | 75 | 81 | 78
  Nausea Grade 1 | 53 | 56 | 54
  Nausea Grade 2 | 16 | 19 | 18
  Nausea Grade 3 | 6 | 6 | 6
  Any Related Nausea | 73 | 73 | 67
  Any Fatigue | 140 | 171 | 171
  Fatigue Grade 1 | 82 | 111 | 99
  Fatigue Grade 2 | 43 | 47 | 58
  Fatigue Grade 3 | 15 | 13 | 14
  Any Related Fatigue | 135 | 163 | 161
  Any Chills | 58 | 54 | 57
  Chills Grade 1 | 43 | 28 | 38
  Chills Grade 2 | 10 | 22 | 13
  Chills Grade 3 | 5 | 4 | 6
  Any Related Chills | 55 | 50 | 53

13. Secondary Outcome: Duration of Solicited General AEs (Pyrexia [Body Temperature Increase], Headache, Myalgia, Nausea, Fatigue and Chills)
Description: Number of days from the start of the general event to resolution. If a participant experienced the general event after both vaccinations, the longer duration is presented. Subjects who had a missing resolution date for the event are not included in the analysis.
Time Frame: as for outcome 11
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
Number analyzed (Participants) | 377 | 375 | 377
Days
  Pyrexia: number analyzed (Participants) | 47 | 60 | 63
  Pyrexia | 2.3 (1.87) | 1.9 (1.91) | 1.9 (1.92)
  Headache: number analyzed (Participants) | 146 | 157 | 155
  Headache | 3.2 (2.85) | 3.1 (2.49) | 3.2 (3.59)
  Myalgia: number analyzed (Participants) | 166 | 173 | 175
  Myalgia | 4.1 (2.8) | 4 (3.27) | 4.1 (3.3)
  Nausea: number analyzed (Participants) | 75 | 81 | 78
  Nausea | 2.6 (2.98) | 2.7 (2.76) | 2.7 (2.5)
  Fatigue: number analyzed (Participants) | 140 | 171 | 171
  Fatigue | 3.9 (5.16) | 3.1 (2.7) | 3.6 (3.57)
  Chills: number analyzed (Participants) | 58 | 54 | 57
  Chills | 2.3 (2.01) | 2.3 (2.71) | 2.3 (2.19)

ADVERSE EVENTS:
Time Frame: Overall study, ie, from first vaccination at Visit 1 through the Follow-up Visit approximately 32 weeks post first vaccination.
Description: Non-systematic assessments include unsolicited adverse events collected at each visit. Systematic events include solicited adverse events collected in a memory aid for 8 days after the vaccinations at Visit 1 (Days 1-8) and Visit 3 (Days 28-35).
Arm/Group | GP 1: Two Doses of FD MVA-BN--Lot 1 | GP 2: Two Doses of FD MVA-BN--Lot 2 | GP 3: Two Doses of FD MVA-BN--Lot 3
All-Cause Mortality (participants affected / at risk) | 0/377 | 2/375 | 0/377
Serious Adverse Events (participants affected / at risk) | 1/377 | 7/375 | 1/377
Other Adverse Events (participants affected / at risk) | 347/377 | 353/375 | 349/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP 1: Two Doses of FD MVA-BN--Lot 1 (N=377) | GP 2: Two Doses of FD MVA-BN--Lot 2 (N=375) | GP 3: Two Doses of FD MVA-BN--Lot 3 (N=377)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0) — Including death during follow-up
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — From follow-up
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — From follow-up
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — From follow-up
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP 1: Two Doses of FD MVA-BN--Lot 1 (N=377) | GP 2: Two Doses of FD MVA-BN--Lot 2 (N=375) | GP 3: Two Doses of FD MVA-BN--Lot 3 (N=377)
Upper respiratory tract infection (Infections and infestations) | 19 (19) | 25 (26) | 21 (23)
Nausea (Gastrointestinal disorders) | 75 (90) | 81 (104) | 78 (96)
Chills (General disorders) | 58 (65) | 54 (62) | 57 (63)
Fatigue (General disorders) | 140 (186) | 171 (225) | 171 (235)
Injection site erythema (General disorders) | 271 (439) | 283 (465) | 272 (459)
Injection site induration (General disorders) | 215 (328) | 226 (355) | 229 (346)
Injection site pain (General disorders) | 325 (573) | 330 (581) | 329 (576)
Injection site pruritis (General disorders) | 210 (303) | 230 (338) | 198 (284)
Injection site swelling (General disorders) | 215 (324) | 233 (343) | 236 (360)
Pyrexia (General disorders) | 47 (56) | 60 (75) | 63 (72)
Myalgia (Musculoskeletal and connective tissue disorders) | 166 (225) | 173 (238) | 175 (241)
Headache (Nervous system disorders) | 146 (189) | 157 (208) | 155 (208)

LIMITATIONS AND CAVEATS:
There were no limitations on the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement entitles Bavarian Nordic to request the Institution(s) to delay their publication for a period of up to six (6) months from the date of the first submission to Bavarian Nordic.

DOCUMENTS (2):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03699124/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03699124/SAP_001.pdf